CLINICAL TRIAL: NCT05796115
Title: PROcalcitonin and Presepsin-guided Decision for Antibiotic Prophylaxis of Early-Onset SEpsis in Preterm Infants: a Multicentre, Randomised Controlled Trial
Brief Title: PROcalcitonin and Presepsin-guided Decision for Antibiotic Prophylaxis of EOS
Acronym: PROPOSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Carlo Dani, Full Professor of Pediatrics, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PROPOSE02
Record Dates: First submitted 2023-03-08; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Early-Onset Neonatal Sepsis
Keywords: Early-Onset Sepsis; Procalcitonin; Presepsin; Preterm infant
MeSH Terms: conditions — Neonatal Sepsis; Premature Birth | interventions — Procalcitonin; Antibiotic Prophylaxis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotic prophylaxis for EOS (Active Comparator)
  Interventions: Procedure: Antibiotic prophylaxis for EOS
- Procalcitonin/Presepsin guided antibiotic prophylaxis for EOS (Experimental)
  Interventions: Procedure: Procalcitonin/Presepsin guided antibiotic prophylaxis for EOS

INTERVENTIONS:
Procedure: Procalcitonin/Presepsin guided antibiotic prophylaxis for EOS — Infants will receive antibiotic prophylaxis for EOS on the basis of Procalcitonin and Presepsin values measured within the first 3 hours of life.
  Arms: Procalcitonin/Presepsin guided antibiotic prophylaxis for EOS
Procedure: Antibiotic prophylaxis for EOS — Infants will receive antibiotic prophylaxis for EOS.
  Arms: Antibiotic prophylaxis for EOS

SUMMARY:
The goal of this randomized controlled study is to compare the outcome of preterm infants who will receive the standard antibiotic prophylaxis for EOS or Procalcitonin/Presepsin-guided antibiotic prophylaxis of early onset sepsis (EOS).

The main question it aims to answer is:

• Does Procalcitonin/Presepsin-guided antibiotic prophylaxis of (EOS) increase survival without major morbidities, including IVH >3 grade, PVL, ROP >3 grade in either eye, NEC >2 grade, BPD, or LOS.

Infants with gestational age between 25+0 and 31+6 weeks of gestation or a birth weight <1500 g will be eligible for enrollment in the study.

Participants will be randomized to receive standard antibiotic prophylaxis for EOS (standard group) or to receive antibiotic prophylaxis for EOS on the basis of PCT/P-SEP measured within 3 h of life (intervention group).

ELIGIBILITY:
Inclusion Criteria:

* infants of 25+0- 31+6 weeks of gestational age will be enrolled in the study.

Exclusion Criteria:

* Risk factors for EOS:

  * maternal GBS colonization without adequate prophylaxis;
  * clinical chorioamnionitis diagnosed by maternal intrapartum fever (either a single documented maternal intrapartum temperature of ≥39.0°C or a temperature of 38.0-38.9°C that persists for >30 minutes) and 1 or more of the following: (1) maternal leukocytosis, (2) purulent cervical drainage, and (3) fetal tachycardia;
  * pre-labor rupture of membranes (ROM) >1 h before delivery.
* Surgery within the first week of life,
* major congenital malformations,
* chromosomal syndromes,
* inherited metabolic disorders,
* fetal hydrops

Ages: 0 Hours to 3 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 266 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Survival without major morbidities. | Participants will be monitored for the duration of hospital stay which is an average of 10 weeks
  Survival without IVH >/=3 grade, PVL, ROP >3 grade in either eye, NEC >2 grade, BPD, or LOS.

SECONDARY OUTCOMES:
Individual components of the composite primary outcome will be regarded as secondary outcomes. | Participants will be monitored for the duration of hospital stay which is an average of 10 weeks
  Occurrence of IVH >/=3 grade, PVL, ROP >3 grade in either eye, NEC >2 grade, BPD, or LOS.

IPD SHARING:
Plan to Share IPD: Undecided